CLINICAL TRIAL: NCT06276049
Title: Enhancement of Self-Directed Learning Through Custom GPT's AI Facilitation Among Medical Students: A Open-label, Randomized Controlled Trial
Brief Title: ChatGPT Helping Advance Training for Medical Students: A Study on Self-Directed Learning Enhancement
Acronym: CHAT-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wang Shalong (Other)
Collaborators: Central South University (Other)
Responsible Party: Sponsor-Investigator, Wang Shalong, Attending Physician of Geriatric Surgery, Central South University
Organization: Central South University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: DGETRRP2023-54
Record Dates: First submitted 2024-02-17; First posted 2024-02-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Self-Directed Learning; Artificial Intelligence; Medical Education
Keywords: self-directed learning; Artificial Intelligence; Medical Education; ChatGPT; large language model

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Engage in 12 weeks of SDL task-based training with LearnGuide's support.
  Interventions: Other: custom GPT supported self-directed learning
- control group (No Intervention): the control group engaged in SDL task-based training without the support of LearnGuide or any similar artificial intelligence (AI) assistance.

INTERVENTIONS:
Other: custom GPT supported self-directed learning — The intervention in our study involved a LearnGuide utilization guide course along with a 12-week integrated training program that incorporated LearnGuide. In the first two-hour session, instructional staff introduced LearnGuide through a hands-on demonstration, teaching students how to use ChatGPT effectively by crafting high-quality prompts. The team emphasized LearnGuide's role as an "AI facilitator" in self-directed learning (SDL). Following the introduction, students were assigned various tasks including online learning, literature reviews, case analyses, and Problem-Based Learning (PBL) activities. Over the 12-week SDL phase with LearnGuide, students were required to complete at least one of these tasks weekly. This setup allowed students to consult mentors for any LearnGuide-related questions, enhancing their learning experience.
  Arms: Intervention group

SUMMARY:
The goal of this clinical trial is to evaluate the effect of LearnGuide, a custom GPT developed with ChatGPT for supporting self-directed learning (SDL) in medical students. The main questions it aims to answer are:

How does LearnGuide influence SDL skills among medical students? Can LearnGuide improve critical thinking and learning flow as measured by Cornell Critical Thinking Test (CCTT) Level Z score and Global Flow Score (GFS)?

Participants will:

Undergo a two-hour introduction to LearnGuide. Engage in 12 weeks of SDL task-based training with LearnGuide's support.

If there is a comparison group: Researchers will compare the group utilizing LearnGuide for SDL and the group without this tool to see if there is a significant difference in SDL skills, critical thinking, and learning flow experiences.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate and postgraduate students studying at the Second Xiangya Hospital
* with access to ChatGPT

Exclusion Criteria:

* utilization of large language models for learning assistance more than once weekly for a period exceeding 2 months.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2023-11-25 (Actual); Primary Completion 2024-03-18 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Self-Directed Learning Scale | at 6 ，12 and 14 weeks
  Utilizing a five-point Likert scale across ten items, assesses learning autonomy in adolescents and adults. Anchored in Brockett's framework, it quantifies learners' independent learning inclination, exhibiting robust internal consistency and validity

SECONDARY OUTCOMES:
Cornell Critical Thinking Test (CCTT) Level Z | at 6 ，12 and 14 weeks
  The CCTT Level Z measures cognitive abilities in students beyond 11th grade with 52 multiple-choice questions across six domains based on the Ennis and Millman Theory, including deductive and inductive reasoning, semantic analysis, credibility assessment, experimental planning, and assumption identification
Flow Short Scale | at 6 and 12 weeks
  The Flow Short Scale (FSS), a condensed form of the Flow State Scale, features ten items on a 7-point scale to assess the flow experience across various activities, from sports to gaming. Its concise yet comprehensive format has made it widely used for evaluating flow experiences in diverse settings

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Geriatirc Surgery, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided
In our study, the decision regarding the sharing of individual participant data (IPD) has not yet been made due to ongoing considerations about privacy, consent, and data protection. We are currently evaluating the ethical implications and ensuring compliance with relevant data protection regulations before making a decision. Additionally, we aim to assess the feasibility of anonymizing IPD in a manner that maintains the integrity and utility of the data for potential future research. Our priority is to safeguard participant confidentiality and respect their consent preferences, while also considering the value of data sharing for advancing scientific knowledge. Further discussions and consultations with stakeholders are planned to reach a well-informed decision.

REFERENCES:
- [Derived] Shalong W, Yi Z, Bin Z, Ganglei L, Jinyu Z, Yanwen Z, Zequn Z, Lianwen Y, Feng R. Enhancing self-directed learning with custom GPT AI facilitation among medical students: A randomized controlled trial. Med Teach. 2025 Jul;47(7):1126-1133. doi: 10.1080/0142159X.2024.2413023. Epub 2024 Oct 19. PMID 39425996